CLINICAL TRIAL: NCT01566253
Title: Comparison of a Patient Controlled Oral Administration (PCOA) of Analgesic Protocol With an IV Administration After Planned Caesarian Section : Monocentric, Randomised and Controlled Study
Brief Title: Oral Self Medication Versus IV Administration of Pain Killers After Caesarian Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Club anesthésie Reanimation Obstetricale (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8832; 2011-004919-23 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Caesarian Section
Keywords: planned caesarian section, analgesic, PCOA
MeSH Terms: interventions — Acetaminophen; Ketoprofen; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCOA (Experimental): The PCOA arm receiving oral self administered multimodal analgesic protocol (paracetamol, ketoprofen, morphine) by oral use.
  Interventions: Drug: Acetaminophen, ketoprofen, morphine
- Standard/ IV (Active Comparator): The standard/IV arm will be received the analgesic treatment by intravenous use, administered by nursing staff.
  Interventions: Drug: Acetaminophen, ketoprofen,morphine

INTERVENTIONS:
Drug: Acetaminophen, ketoprofen, morphine — Acetaminophen 0.5g, maximum 4g by day, 48 hours ketoprofen 100 mg, twice a day, 48 hours Morphine 10 mg, maximum 90 mg by day, 36 hours
  Other Names: dolipraneoro 500mg, MA 352 120-2; bi profenid LP 100 mg, MA 399804-5; Actiskenan 10 mg, MA 561958-9
  Arms: PCOA
Drug: Acetaminophen, ketoprofen,morphine — Acetaminophen 1g/100 ml IV, maximum 4g by 24 hours, 48 hours Ketoprofen IV, maximum 0,2 gram by 24 hours, 48 hours Morphine IV,maximum 60mg by 24 hours, 36 hours.
  Other Names: Paracetamol 1g/100 ml IV : MA #571860-1; Profenid IV : MA #557466-8; Morphine IV : MA #566945-2
  Arms: Standard/ IV

SUMMARY:
C-section deliveries are painful and need adequate analgesia. In the same time, mothers need early rehabilitation to take care of the baby.

Hypothesis: Early oral self administration of painkillers could be as effective as usual IV administration by nursing staff.

Purpose of the study: Evaluation of the efficacy of a program of self administration of painkillers postoperatively of C-section delivery.

DETAILED DESCRIPTION:
Two Arms: PCOA group receiving oral self administered multimodal analgesic protocol and IV group receiving same multimodal analgesic protocol administered by nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* planned caesarian section

Exclusion Criteria:

* delivery bleeding which requires general anaesthetic and other surgical treatment
* contraindication of the targetted anaesthetic because of hemostatis dysfunctionments
* Signed consent form
* under 18 years old, toxicomania
* do not french speacking
* allergia or contraindication to IMPs
* suffer from chronicle disease
* do not affiliate to a health protection
* do not want to cooperate with the medical staff

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Median pain score during the first 48 hours (Verbal rating PAin Scale) | After 48 hours
  The pain score will be assessed by investigators at different times : H2 (2 hours after the end of the caesarian), H6, H12, H18, H24, H30, H36 and H48.

SECONDARY OUTCOMES:
Onset of the first request of rescue analgesic drug | maximum 48 hours following the caesarian
  If the study analgesic treatment is not enough, a rescue analgesic drug could administered by nursing staff.

CONTACTS AND LOCATIONS:
Overall Officials: Estelle Morau, Doctor, Principal Investigator — University Hosptial of Montpellier
Locations (1):
- university Hospital, Arnaud de Villeneuve, Gynecology department, Montpellier, France